CLINICAL TRIAL: NCT04142827
Title: The Effect of Long Term Therapy With High Flow Humidification Compared to Usual Care
Brief Title: The Effect of Long Term Therapy With High Flow Humidification Compared to Usual Care in Patients With Bronchiectasis (BX)
Acronym: BX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Giuseppe Fiorentino (Other)
Responsible Party: Sponsor-Investigator, Dr. Giuseppe Fiorentino, Director Giuseppe Fiorentino, Monaldi Hospital
Organization: Monaldi Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: High Flow in Bronchiectasis
Record Dates: First submitted 2019-10-21; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Bronchiectasis Adult; Lung Infection; Quality of Life; Humidifier Lung; COPD Exacerbation; COPD Asthma
Keywords: Bronchiectasis; High Flow Therapy; Humidifcation; Lung Infection; Quality of life
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy with high flow humidification (Experimental): The patients will be activated after enrollment with myAirvo2 device at home for 6 months before first observations
  Interventions: Device: High Flow Humidification
- Therapy with usual care (No Intervention): The patients will be under usual care for observational

INTERVENTIONS:
Device: High Flow Humidification — myAirvo2 gives at home for long therapy treatment
  Arms: Therapy with high flow humidification

SUMMARY:
The study is intended to understand the benefit of Long Term Home care Therapy with nasal High flow in Bronchiectasis patients at home. Primary end point is to evaluate daily life compared to usual care and secondary is to evaluate the changes in lung function

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Bronchiectasis on HRCT
* Optimization of Therapy for at least 15 days before enrollment
* Autonomous patients with possibilities of practicing rehabilitations cycles

Exclusion Criteria:

* OSAS (ODI>10/h)
* HOME NIV
* PH<7,35 - paO2< 60mmHg, paCo2> 55 mmHg
* Lung cancer
* Contraindication to high-flow nasal cannula (hfnc)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-03-03 (Estimated); Study Completion 2020-09-03 (Estimated)

PRIMARY OUTCOMES:
Improvment Daily Life | 1 year
  measurement via questionary SGRQ
measurement of Sputum production | 1 year
  Microbiological Mesurement of sputum
measurement Exercise tolerance | 1 year
  measurement with 6 minutes walking test
Number of missed working or school day | 1 year
  Calculation of days of sick
time from first exacerbations | 1 year
  measurement of time dalay from last exacerbation
number of exacerbations including their durations and severity | 1 year
  counting form their clinic diary of number of exacerbation

SECONDARY OUTCOMES:
Evaluation of Arterial Blood Glass | 1 year
  Arterial Blood Glass draw at time zero and time 1
Unit of Nitric Oxide | 1 year
  Measurement with Nitric oxide device
Evaluation of Reactive C-Protein | 1 year
  comparation of blood draw

CONTACTS AND LOCATIONS:
Locations (1):
- Rosa Cauteruccio, Napoli, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol